CLINICAL TRIAL: NCT01137760
Title: Protocol 1: Galactooligosaccharide, Immune Strength, and Digestive Health in Academically Stressed University Students
Brief Title: Galactooligosaccharide, Immune Strength, and Digestive Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: GTC Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 307-2009
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: adults; fiber; cold; flu; stress; microbiota
MeSH Terms: conditions — Common Cold; Influenza, Human | interventions — Sucrose; 4'-galactooligosaccharide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sugar pill (Placebo Comparator)
  Interventions: Dietary Supplement: Sucrose
- Galactooligosaccharide 2.5 g (Experimental)
  Interventions: Dietary Supplement: Galactooligosaccharide
- Galactooligosaccharide 5.0 g (Experimental)
  Interventions: Dietary Supplement: Galactooligosaccharide

INTERVENTIONS:
Dietary Supplement: Sucrose — 5 g of sucrose daily for 8 weeks
  Arms: Sugar pill
Dietary Supplement: Galactooligosaccharide — 2.5 g galactooligosaccharide plus 2.5 g sucrose daily for 8 weeks
  Arms: Galactooligosaccharide 2.5 g
Dietary Supplement: Galactooligosaccharide — 5.0 g galactooligosaccharide daily for 8 weeks
  Arms: Galactooligosaccharide 5.0 g

SUMMARY:
The purpose of this research study is to determine whether a functional fiber, galactooligosaccharide, can help maintain immune strength and digestive health in undergraduate students who are undergoing an academic stress (i.e., final exams). Subjects will be asked to consume the fiber or placebo each day for eight weeks. Immune and gastrointestinal health will be evaluated via daily questionnaires obtained from 420 students and from the collection of fecal samples in a subgroup of students.

DETAILED DESCRIPTION:
A prospective, randomized, parallel, double-blind, placebo controlled design will be used. Healthy full-time undergraduate students undergoing fall 2009 final academic exams will be recruited from the University of Florida. Informed consent will be obtained. All subjects will be consented for the main intervention study and a subgroup (n=25/group or 75 total) of these subjects will also be consented to provide two stool samples at baseline and two stool samples during the week of final exams (approximately week 4 of the intervention). Subjects will be stratified based on gender and randomized (n=140/group) to receive 0 g, 2.5 g, or 5.0 g of the fermentable fiber, galactooligosaccharides, for eight weeks around the time of their fall final exams. Subjects will complete daily online questionnaires asking whether they are experiencing any cold/flu symptoms. Weekly online questionnaires will collect information regarding gastrointestinal symptoms over the past week. The acute psychological stress associated with final exams will increase cold/flu symptoms. It is anticipated that students consuming the galactooligosaccharides versus the placebo will have more healthy days (i.e., days without cold symptoms) due to fiber induced changes in the beneficial bacteria within the colon, which reduces the burden on the immune system.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* willing to complete a daily assessment form via computer
* willing to discontinue any immune-enhancing dietary supplements ( e.g., prebiotics and fiber supplements, probiotics, echinacea, fish oil, vitamin E >100% of the RDA or >15 mg/day)
* willing to take the fiber for 8 weeks
* had a cold in last 12 months
* have at least 1 final during the Fall 2009 exam week, between Saturday, December 12 and Friday, December18, 2009
* daily access to a computer with Internet access for the entire 8-wk study

Exclusion Criteria:

* current smoker
* chronic allergies involving the upper respiratory tract (Chronic = taking allergy medicine daily)
* an allergy to milk
* known illnesses or conditions that may impact perceived health such as HIV/AIDS, diabetes, renal or gastrointestinal diseases
* received chemotherapy or other immune suppressing therapy within the last year
* antibiotic therapy in the past two months
* a cold or cold symptoms (on day of randomization)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Days without cold/flu symptoms | Measured daily for 8 weeks
  Number of cold/flu symptoms (running/congested nose, stiffness or chills, headache, cough, fatigue, fever, sore throat, achiness, ear discomfort), Intensity of cold/flu symptoms

SECONDARY OUTCOMES:
Gastrointestinal symptoms | Measured weekly for 8 weeks
  diarrhea, loose stools, urgent need for defecation, rumbling, bloating, burping, gas, constipation, hard stools, feeling of incomplete evacuation, abdominal pain, hunger pains, nausea, heartburn, acid regurgitation
Changes in overall microbiota diversity | Measured at baseline and approximately week 4
  Stool collections will be obtained from a subgroup of subjects (n=25/group or 75 total). Samples will be provided at baseline (i.e., before the start of the intervention)and during the week of final exams (i.e., approximately study week 4).

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, PhD, RD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Result] Hughes C, Davoodi-Semiromi Y, Colee JC, Culpepper T, Dahl WJ, Mai V, Christman MC, Langkamp-Henken B. Galactooligosaccharide supplementation reduces stress-induced gastrointestinal dysfunction and days of cold or flu: a randomized, double-blind, controlled trial in healthy university students. Am J Clin Nutr. 2011 Jun;93(6):1305-11. doi: 10.3945/ajcn.111.014126. Epub 2011 Apr 27. PMID 21525194